CLINICAL TRIAL: NCT04632030
Title: Shrinking the Size of the Tobacco Power Wall and Restricting the Number of Tobacco Products Displayed to Reduce Adolescent Tobacco Use
Brief Title: Shrinking the Size of the Tobacco Power Wall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, William Shadel, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA050972 (NIH)
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): The tobacco power wall and number of products appears in a typical format: large power wall with a large number of products (defined here as three large cabinets)
  Interventions: Behavioral: Tobacco power wall size and tobacco products displayed
- Small (Experimental): The tobacco power wall and number of tobacco products appear in their smallest format: small power wall with a small number of products displayed (defined here as one large cabinet)
  Interventions: Behavioral: Tobacco power wall size and tobacco products displayed
- Medium (Experimental): The tobacco power wall and number of tobacco products appear in a format sized between the control and small conditions: a medium sized power wall with a medium number of products displayed (defined here as two large cabinets).
  Interventions: Behavioral: Tobacco power wall size and tobacco products displayed

INTERVENTIONS:
Behavioral: Tobacco power wall size and tobacco products displayed — The intervention varies the size of the tobacco power wall and number of tobacco products displayed on it.

SUMMARY:
The overall aim of this research is to experimentally evaluate the extent to which reducing the size of the tobacco power wall and the number of tobacco product units displayed influences tobacco use risk in adolescents.

DETAILED DESCRIPTION:
This experiment will take place in the RAND StoreLab (RSL), a life-sized replica of a convenience store that we developed to evaluate how altering aspects of tobacco promotion at POS influences tobacco use risk during simulated shopping experiences. The study will use a between-subjects design, in which adolescents are randomly assigned to shop in the RSL under one of three conditions: (1) Large power wall/ multiple product units displayed; (2) Medium-sized power wall/multiple product units displayed; and (3) Small power wall/single product units displayed. We will consider the effect of these power wall alterations on risk of use of four classes of tobacco products: cigarettes, electronic nicotine delivery devices, cigarillos, and smokeless tobacco.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 11 and 20

Exclusion Criteria:

* any medical or psychological condition that would make participation in the procedures of the study difficult (based on self-report).

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 275 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RAND, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Small | Medium
Started | 96 | 86 | 93
Completed | 96 | 86 | 93
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Small | Medium | Total
Number analyzed (Participants) | 96 | 86 | 93 | 275
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (3.2) | 16.6 (3.1) | 16.4 (3.0) | 16.6 (3.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 26 | 26 | 30 | 82
  Female | 65 | 55 | 58 | 178
  Nonbinary/other | 5 | 5 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 3 | 12
  Not Hispanic or Latino | 90 | 82 | 90 | 262
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 13 | 9 | 21 | 43
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 7 | 20
  White | 66 | 64 | 55 | 185
  More than one race | 7 | 4 | 7 | 18
  Unknown or Not Reported | 3 | 1 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 96 | 86 | 93 | 275

OUTCOME MEASURES:

1. Primary Outcome: Proportion at Risk for Cigarette Smoking
Description: A two item self-report assessment: 1) If one of your best friends offered you an unflavored cigarette would you use it? 2) If one of your best friends offered you a menthol cigarette would you use it? Responses to each item are made on a 10-point scale where 1 = definitely not; and 10 = definitely yes and responses across the two items are summed for a total scale score. Total scale scores are dichotomized: scores of 2 are coded as '0' (no risk) and any score greater than 2 is coded as '1' (at risk). Outcome is proportion at risk of cigarette smoking (number of participants at risk over number of participants within condition).
Time Frame: within 5 minutes of the intervention
Population: Sample size may differ from baseline because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Control | Small | Medium
Number analyzed (Participants) | 82 | 80 | 78
proportion of participants | .18 [.11 to .29] | .39 [.27 to .53] | .26 [.16 to .38]
Statistical Analysis 1: Comparison: Control vs Medium; Test type: Other; Odds Ratio (OR) = 1.58, 95% CI 2-sided [.69 to 3.6] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Control vs Small; Test type: Other; Odds Ratio (OR) = 2.89, 95% CI 2-sided [1.28 to 6.55] — Adjusted for age, education, and lifetime tobacco use

2. Primary Outcome: Proportion at Risk of Using Electronic Nicotine Delivery Devices (ENDS)
Description: A three item, self-report assessment: 1) If one of your best friends offered you an unflavored vaping product would you use it? 2) If one of your best friends offered you a vaping product flavored with menthol or mint, would you use it? 3) If one of your best friends offered you a vaping product flavored with fruit, candy, alcohol or non-alcohol drink, or some other sweet flavor, would you use it? Responses to each item are made on a 10-point scale where 1 = definitely not; and 10 = definitely yes and responses across the three items are summed for a total scale score. Total scale scores are dichotomized: scores of 3 are coded as '0' (no risk) and any score greater than 3 is coded as '1' (at risk). Outcome is proportion at risk of ENDS use (number of participants at risk over number of participants within condition).
Time Frame: within 5 minutes of the intervention
Population: Sample sizes may differ from baseline because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Control | Small | Medium
Number analyzed (Participants) | 81 | 78 | 81
proportion of participants | .34 [.22 to .47] | .59 [.46 to .72] | .59 [.45 to .72]
Statistical Analysis 1: Comparison: Control vs Medium; Test type: Other; Odds Ratio (OR) = 2.88, 95% CI 2-sided [1.28 to 6.47] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Control vs Small; Test type: Other; Odds Ratio (OR) = 2.87, 95% CI 2-sided [1.26 to 6.50] — Adjusted for age, education, and lifetime tobacco use

3. Primary Outcome: Proportion at Risk of Using Smokeless Tobacco
Description: A three item self report assessment: : 1) If one of your best friends offered you unflavored smokeless tobacco would you use it? 2) If one of your best friends offered you smokeless tobacco flavored with flavored with menthol, mint, spearmint, or wintergreen would you use it? 3) If one of your best friends offered you smokeless tobacco flavored with fruit would you use it? Responses to each item are made on a 10-point scale where 1 = definitely not; and 10 = definitely yes and responses across the three items are summed for a total scale score. Total scale scores are dichotomized: scores of 3 are coded as '0' (no risk) and any score greater than 3 is coded as '1' (at risk).Outcome is proportion at risk of smokeless tobacco use (number of participants at risk over number of participants within condition).
Time Frame: within 5 minutes of the intervention
Population: Sample size may differ from baseline due to missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Control | Small | Medium
Number analyzed (Participants) | 81 | 77 | 78
proportion of participants | .12 [.06 to .21] | .20 [.12 to .31] | .17 [.10 to .27]
Statistical Analysis 1: Comparison: Control vs Medium; Test type: Other; Odds Ratio (OR) = 1.51, 95% CI 2-sided [.59 to 3.86] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Control vs Small; Test type: Other; Odds Ratio (OR) = 1.85, 95% CI 2-sided [.73 to 4.67] — Adjusted for age, education, and lifetime tobacco use

4. Primary Outcome: Proportion at Risk of Using Little Cigar/Cigarillos (LCC)
Description: A three item, self report assessment: 1) If one of your best friends offered you an unflavored cigarillos/filtered cigar would you use it? 2) If one of your best friends offered you a cigarillos/filtered cigar flavored with menthol or mint would you use it? 3) If one of your best friends offered you a cigarillos/filtered cigar flavored with fruit, candy, alcohol, or some other sweet flavor, would you use it? Responses to each item are made on a 10-point scale where 1 = definitely not; and 10 = definitely yes and responses across the three items are summed for a total scale score. Total scale scores are dichotomized: scores of 3 are coded as '0' (no risk) and any score greater than 3 is coded as '1' (at risk). Outcome is proportion at risk of LCC use (number of participants at risk over number of participants within condition).
Time Frame: within 5 minutes of the intervention
Population: Sample sizes may differ from baseline due to missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Control | Small | Medium
Number analyzed (Participants) | 80 | 77 | 77
proportion of participants | .17 [.10 to .27] | .31 [.20 to .44] | .20 [.12 to .32]
Statistical Analysis 1: Comparison: Control vs Medium; Test type: Other; Odds Ratio (OR) = 1.25, 95% CI 2-sided [.53 to 2.99] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Control vs Small; Test type: Other; Odds Ratio (OR) = 2.19, 95% CI 2-sided [.94 to 5.13] — Adjusted for age, education, and lifetime tobacco use

ADVERSE EVENTS:
Time Frame: One day
Arm/Group | Control | Small | Medium
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/86 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/86 | 0/93
Other Adverse Events (participants affected / at risk) | 0/96 | 0/86 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT04632030/Prot_SAP_000.pdf